CLINICAL TRIAL: NCT03745677
Title: Redesigning Systems to Improve Quality for Hospitalized Patients
Acronym: RESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Society of Hospital Medicine (Other); University of Michigan (Other); University of Kentucky (Other); The University of Texas Health Science Center at San Antonio (Other); Alamance Regional Medical Center (Unknown); Baptist Hospital (Unknown); Good Samaritan Regional Medical Center, Oregon (Other); Ball Memorial Hospital (Other); University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Kevin O'Leary, Chief, Division of Hospital Medicine, Northwestern University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R18HS025649 (AHRQ)
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Interdisciplinary Communication; Interpersonal Relations; Adverse Event; Interprofessional Relations
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Two group pretest-posttest analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): Each study site has selected 1-2 units ideally suited for initial implementation of the Advanced and Integrated MicroSystems (AIMS) interventions (Phase I Implementation) and 1-2 units for later implementation of AIMS interventions (Phase II Implementation). During Implementation Phase I, AIMS interventions were implemented on the initial, phase I Implementation units. The phase II units serve as control units during phase I.
  Interventions: Behavioral: Advanced and Integrated MicroSystems (AIMS) interventions
- Phase II (Experimental): During Implementation Phase II, Advanced and Integrated MicroSystems (AIMS) interventions are being implemented on additional, phase II implementation units, leveraging lessons learned during phase I.
  Interventions: Behavioral: Advanced and Integrated MicroSystems (AIMS) interventions

INTERVENTIONS:
Behavioral: Advanced and Integrated MicroSystems (AIMS) interventions — Each of 4 sites is receiving mentorship from nurse and physician with expertise in implementing similar interventions. The AIMS interventions consist of 1) unit-based physician teams, 2) unit nurse-physician co-leadership, 3) enhanced interprofessional rounds, 4) unit-level performance reports, and 5) patient engagement activities.

SUMMARY:
Despite recent improvements, healthcare systems are still a long way from consistently delivering high quality care to hospitalized patients. In this study, the research team is assisting hospitals in implementing a set of complementary, mutually reinforcing interventions to redesign care for hospitalized medical patients. The investigators anticipate the interventions will improve teamwork and patient outcomes and that identifiable factors and strategies will be associated with successful implementation.

DETAILED DESCRIPTION:
Most adults requiring hospitalization are admitted for medical conditions, yet the optimal model of care for these patients is yet to be established. Current care delivery models lack the ability to optimally coordinate care on a daily basis and improve performance over time. A growing body of research has tested interventions to redesign aspects of care delivery for hospitalized medical patients. These interventions improve processes and culture, but the evidence that patient outcomes have improved is equivocal. Importantly, most studies have examined the effect of single interventions in isolation, yet these interventions are better conceptualized as complementary and mutually reinforcing components of a redesigned clinical microsystem. Clinical microsystems are the front line care giving units where patients, families, and care teams meet. Our research team developed a set of complementary, mutually reinforcing interventions based on available evidence and anchored in a clinical microsystem framework. The 5 Advanced and Integrated MicroSystems (AIMS) interventions include: 1) Unit-based Physician Teams, 2) Unit Nurse-Physician Co-leadership, 3) Enhanced Interdisciplinary Rounds, 4) Unit-level Performance Reports, 5) Patient Engagement Activities. Our long term goal is to discover and disseminate the optimal model of care to improve outcomes for hospitalized patients. Our specific objective for this proposal is to implement a set of evidence-based complementary interventions across a range of clinical microsystems, identify factors and strategies associated with successful implementation, and evaluate the impact on quality. Our research team is using mentored implementation, i.e., coaching by external professionals who are experts in the area of focus, to help facilitate change. The research team has enrolled 4 hospitals in this quality improvement mentored implementation study. Our hypothesis is that uptake of the complementary components of the intervention set will result in improvements in teamwork climate and patient outcomes.

Specific Aims of the Redesigning Systems to Improve Quality for Hospitalized Patients (RESET) study include:

1. Conduct a multi-site mentored implementation study in which each site adapts and implements complementary interventions to improve care for medical patients.
2. Evaluate the effect of the intervention set on teamwork climate and patient outcomes related to safety, patient experience, and efficiency.
3. Assess how site-specific contextual factors interact with the variation in the intensity and fidelity of implementation to effect teamwork and patient outcomes.

The findings generated from this study will be directly applicable to hospitals throughout the U.S. and our partnership with the Society of Hospital Medicine, the American Nurses Association, and the Institute for Patient- and Family-Centered Care will ensure effective dissemination and impact.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted, under inpatient or observation status, to study units

Exclusion Criteria:

* Patients transferred from other hospitals and those initially admitted to other units.
* Patients admitted under non-medical services on the study units.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4265 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Teamwork climate using the Safety Attitudes Questionnaire (SAQ) | Administered annually in years 1 through 4
  14 item validated survey tool to assess teamwork climate in clinical settings. The survey will be administered via REDcap to all nurses, physicians, pharmacists, social workers, and case managers on study units.
Adverse events | Medical record review of patients hospitalized in years 1 through 3.
  We will use the Medicare Patient Safety Monitoring System (MPSMS) methodology to detect adverse events. MPSMS is a medical record-based national patient safety surveillance system that provides rates for specific inpatient adverse event measures.

SECONDARY OUTCOMES:
Patient experience | Years 1 through 3.
  We will use Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) global ratings of hospital care.
Length of stay | Years 1 through 3
  Length of hospital stay for patients admitted to study unit
30 day readmissions | Years 1 through 3
  30 day readmissions for patients admitted to the study units

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O'Leary, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (4):
- United States (4):
  - Baptist Hospital, Pensacola, Florida
  - Indiana University Ball Memorial Hospital, Muncie, Indiana
  - Alamance Regional Medical Center, Burlington, North Carolina
  - Legacy Good Samaritan Hospital, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Leary KJ, Killarney A, Hansen LO, Jones S, Malladi M, Marks K, M Shah H. Effect of patient-centred bedside rounds on hospitalised patients' decision control, activation and satisfaction with care. BMJ Qual Saf. 2016 Dec;25(12):921-928. doi: 10.1136/bmjqs-2015-004561. Epub 2015 Dec 1. PMID 26628552
- [Background] O'Leary KJ, Creden AJ, Slade ME, Landler MP, Kulkarni N, Lee J, Vozenilek JA, Pfeifer P, Eller S, Wayne DB, Williams MV. Implementation of unit-based interventions to improve teamwork and patient safety on a medical service. Am J Med Qual. 2015 Sep-Oct;30(5):409-16. doi: 10.1177/1062860614538093. Epub 2014 Jun 11. PMID 24919598
- [Background] O'Leary KJ, Buck R, Fligiel HM, Haviley C, Slade ME, Landler MP, Kulkarni N, Hinami K, Lee J, Cohen SE, Williams MV, Wayne DB. Structured interdisciplinary rounds in a medical teaching unit: improving patient safety. Arch Intern Med. 2011 Apr 11;171(7):678-84. doi: 10.1001/archinternmed.2011.128. PMID 21482844
- [Background] O'Leary KJ, Wayne DB, Landler MP, Kulkarni N, Haviley C, Hahn KJ, Jeon J, Englert KM, Williams MV. Impact of localizing physicians to hospital units on nurse-physician communication and agreement on the plan of care. J Gen Intern Med. 2009 Nov;24(11):1223-7. doi: 10.1007/s11606-009-1113-7. Epub 2009 Sep 19. PMID 19768510
- [Background] O'Leary KJ, Johnson JK, Manojlovich M, Astik GJ, Williams MV. Use of Unit-Based Interventions to Improve the Quality of Care for Hospitalized Medical Patients: A National Survey. Jt Comm J Qual Patient Saf. 2017 Nov;43(11):573-579. doi: 10.1016/j.jcjq.2017.05.008. Epub 2017 Jul 21. PMID 29056177
- [Background] Pannick S, Davis R, Ashrafian H, Byrne BE, Beveridge I, Athanasiou T, Wachter RM, Sevdalis N. Effects of Interdisciplinary Team Care Interventions on General Medical Wards: A Systematic Review. JAMA Intern Med. 2015 Aug;175(8):1288-98. doi: 10.1001/jamainternmed.2015.2421. PMID 26076428
- [Background] Singh S, Tarima S, Rana V, Marks DS, Conti M, Idstein K, Biblo LA, Fletcher KE. Impact of localizing general medical teams to a single nursing unit. J Hosp Med. 2012 Sep;7(7):551-6. doi: 10.1002/jhm.1948. Epub 2012 Jul 12. PMID 22791661
- [Background] Nelson EC, Godfrey MM, Batalden PB, Berry SA, Bothe AE Jr, McKinley KE, Melin CN, Muething SE, Moore LG, Wasson JH, Nolan TW. Clinical microsystems, part 1. The building blocks of health systems. Jt Comm J Qual Patient Saf. 2008 Jul;34(7):367-78. doi: 10.1016/s1553-7250(08)34047-1. PMID 18677868
- [Background] Kara A, Johnson CS, Nicley A, Niemeier MR, Hui SL. Redesigning inpatient care: Testing the effectiveness of an accountable care team model. J Hosp Med. 2015 Dec;10(12):773-9. doi: 10.1002/jhm.2432. Epub 2015 Aug 19. PMID 26286828
- [Background] Stein J, Payne C, Methvin A, Bonsall JM, Chadwick L, Clark D, Castle BW, Tong D, Dressler DD. Reorganizing a hospital ward as an accountable care unit. J Hosp Med. 2015 Jan;10(1):36-40. doi: 10.1002/jhm.2284. Epub 2014 Nov 17. PMID 25399928
- [Background] Li J, Hinami K, Hansen LO, Maynard G, Budnitz T, Williams MV. The physician mentored implementation model: a promising quality improvement framework for health care change. Acad Med. 2015 Mar;90(3):303-10. doi: 10.1097/ACM.0000000000000547. PMID 25354069
- [Derived] O'Leary KJ, Johnson JK, Williams MV, Estrella R, Hanrahan K, Leykum LK, Smith GR, Goldstein JD, Kim JS, Thompson S, Terwilliger I, Song J, Lee J, Manojlovich M. Effect of Complementary Interventions to Redesign Care on Teamwork and Quality for Hospitalized Medical Patients : A Pragmatic Controlled Trial. Ann Intern Med. 2023 Nov;176(11):1456-1464. doi: 10.7326/M23-0953. Epub 2023 Oct 31. PMID 37903367
- [Derived] O'Leary KJ, Johnson JK, Manojlovich M, Goldstein JD, Lee J, Williams MV. Redesigning systems to improve teamwork and quality for hospitalized patients (RESET): study protocol evaluating the effect of mentored implementation to redesign clinical microsystems. BMC Health Serv Res. 2019 May 8;19(1):293. doi: 10.1186/s12913-019-4116-z. PMID 31068161